CLINICAL TRIAL: NCT05738772
Title: Diagnostic Accuracy of APAC, ASAP and GALAD Scores in Hepatocellular Carcinoma Among Cirrhotic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Mahmoud Mohammed Mohammed, assistant lecturer, Sohag University
Other Study IDs: Soh-Med-23-02-15
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hcc group: The study group will include 45 patients with HCC on top of liver cirrhosis. All virus-related liver cirrhosis and all BCLC stages of HCC will be accepted. Verified presence of HCC, will be assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) or based on histological validation. In patients with presence of liver cirrhosis, non-invasive diagnosis of HCC is standard, when dynamic imaging shows typical diagnostic patterns as the combination of hypervascularity in late arterial phase and washout on portal venous and/or delayed phases
  Interventions: Diagnostic Test: serum sample for ELIZA
- LC group: Will include 45 patients diagnosed with liver cirrhosis on top of HCV or HBV with an absence of focal lesions on ultrasound screening as a control group. Cirrhosis will be determined according to clinical, serological, and radiological findings
  Interventions: Diagnostic Test: serum sample for ELIZA

INTERVENTIONS:
Diagnostic Test: serum sample for ELIZA — Assay of AFP, AFP-L3, DCP and Soluble PDGFRβwill be done by enzyme-linked immunosorbent assay (ELISA).

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver malignancy with most patients developing HCC due to chronic liver diseases. Unfortunately, HCC has a morality to incidence ratio that approaches 1.

Among the etiological factors associated with HCC, hepatitis C virus (HCV) and Hepatitis B virus (HBV) infections are major risk factors. Despite HBV vaccination programs and effective direct antiviral agents (DAA) for treatment of HCV, the incidence of virus-related HCC remains high. HCV eradication by antiviral treatment reduces but does not eliminate HCC risk. Patients with HCV-related cirrhosis require HCC surveillance even after sustained virologic response (SVR) due to a persistent risk of HCC even years after SVR . In Egypt, HCC represents the fourth common cancer and is the most common cause of mortality-related and morbidity-related cancer. Egypt ranks the third and 15th most populous country in Africa and worldwide, respectively, and the Egyptian health authorities consider HCC as one of the most challenging health problems for the current decade. Both HCC screening and monitoring efforts have improved significantly since 2018 as a result of the national screening campaign .The early diagnosis of HCC is essential to initiate curative treatments to improve short term and long-term prognosis. Therefore, highly effective methods are needed to detect HCC at an earlier stage. American Association for the Study of Liver Diseases (AASLD) and European Association for the Study of the Liver (EASL) guidelines recommend the periodic use of ultrasound scanning (USS), with or without Alpha-fetoprotein (AFP) evaluation, for HCC surveillance. However, suboptimal performance of USS has been reported, with its sensitivity being compromised by the extent of liver cirrhosis, high body mass index (BMI), etiology of liver disease, expertise of the operator and quality of the equipment. Moreover, its sensitivity and specificity for early-stage HCC was found to be rather low . Serum biomarkers play an essential role in diagnosing HCC, as biomarkers are often more convenient, inexpensive, non-invasive, and reproducible . Alpha-fetoprotein (AFP) is a widely used biomarker for HCC diagnosis. The diagnostic accuracy of AFP is limited, however, due to its high false-negative rate to detect small or early stage tumors. As previous studies have demonstrated, the sensitivity of AFP among patients with HCC was 52% for tumors > 3cm and dropped to only 25% for tumors < 3cm. In addition, AFP may also be elevated in some benign liver diseases, such as chronic hepatitis and cirrhosis even in the absence of HCC.

ELIGIBILITY:
Inclusion Criteria:

* A total of 90 adult patients with liver cirrhosis attending the outpatient clinic or inpatient section of the department of tropical medicine and gastroenterology at Sohag University Hospital will be included in the study. Patients will be divided into two groups

Exclusion Criteria:

* 1. patients aged <18 years old. 2. Presence of clinically suspected other causes of hepatocellular injury (any history of alcoholism, autoimmune hepatitis, primary sclerosing cholangitis (PSC), primary biliary cholangitis (PBC), Wilson's disease, fatty liver diseases with metabolic syndrome & drug induced liver disease). 3. Receipt of any tumor specific therapy before blood samples collection. 4. Any patients who are on warfarin will be excluded as warfarin can elevate the DCP level in the absence of HCC. 5. Patients having malignancies other than HCC. 6. Presence of distant metastasis. 7. Presence of venous thromboembolism including portal vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 90 adult patients with liver cirrhosis attending the outpatient clinic or inpatient section of the department of tropical medicine and gastroenterology at Sohag University Hospital will be included in the study. Patients will be divided into two groups.:
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
serum level of AFP-L3. | one year
  Assay of AFP-L3 will be done by enzyme-linked immunosorbent assay (ELISA) then Diagnostic scoring tools were calculated using the following formulae:The GALAD score will be calculated using the following equation: GALAD score = - 10.08 + 0.09 × age + 1.67 × gender + 2.34 × Lg (AFP [ng/ml]) + 0.04 × AFP-L3%% + 1.33 × Lg (PIVKA-II [mAU/ml]), where gender = 0 for females and 1 for males. - The probability of HCC in a patient was calculated as follows: Pr (HCC)=exp (Z)/ (1 + exp (Z)) (z: GALAD)The ASAP score was calculated using the following equation: ASAP score = -7.58 + 0.05
  × age - 0.58 × gender +0.42 × Ln (AFP [ng/ml]) + 1.11 × Ln (PIVIKA-II [mAU/ml]), where gender = 0 for males and 1 for femalesThe APAC score = (Age [years] x 0.20480) - (log10(sPDGFRβ [pg/mL]) x 1.98684) + (log10(AFP [ng/mL]) x 2.45657) - (Creatinine [mg/dL] x 2.46891) - 4.36493
serum level of DCP | 1 year
  Assay of DCP will be done by enzyme-linked immunosorbent assay (ELISA) then Diagnostic scoring tools were calculated using the following formulae:The GALAD score will be calculated using the following equation: GALAD score = - 10.08 + 0.09 × age + 1.67 × gender + 2.34 × Lg (AFP [ng/ml]) + 0.04 × AFP-L3%% + 1.33 × Lg (PIVKA-II [mAU/ml]), where gender = 0 for females and 1 for males. - The probability of HCC in a patient was calculated as follows: Pr (HCC)=exp (Z)/ (1 + exp (Z)) (z: GALAD)The ASAP score was calculated using the following equation: ASAP score = -7.58 + 0.05
  × age - 0.58 × gender +0.42 × Ln (AFP [ng/ml]) + 1.11 × Ln (PIVIKA-II [mAU/ml]), where gender = 0 for males and 1 for femalesThe APAC score = (Age [years] x 0.20480) - (log10(sPDGFRβ [pg/mL]) x 1.98684) + (log10(AFP [ng/mL]) x 2.45657) - (Creatinine [mg/dL] x 2.46891) - 4.36493
Serum level of Soluble PDGFRβ | 1 year
  Assay of Soluble PDGFRβ will be done by enzyme-linked immunosorbent assay (ELISA) then Diagnostic scoring tools were calculated using the following formulae:The GALAD score will be calculated using the following equation: GALAD score = - 10.08 + 0.09 × age + 1.67 × gender + 2.34 × Lg (AFP [ng/ml]) + 0.04 × AFP-L3%% + 1.33 × Lg (PIVKA-II [mAU/ml]), where gender = 0 for females and 1 for males. - The probability of HCC in a patient was calculated as follows: Pr (HCC)=exp (Z)/ (1 + exp (Z)) (z: GALAD)The ASAP score was calculated using the following equation: ASAP score = -7.58 + 0.05
  × age - 0.58 × gender +0.42 × Ln (AFP [ng/ml]) + 1.11 × Ln (PIVIKA-II [mAU/ml]), where gender = 0 for males and 1 for femalesThe APAC score = (Age [years] x 0.20480) - (log10(sPDGFRβ [pg/mL]) x 1.98684) + (log10(AFP [ng/mL]) x 2.45657) - (Creatinine [mg/dL] x 2.46891) - 4.36493

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caviglia GP, Ribaldone DG, Abate ML, Ciancio A, Pellicano R, Smedile A, Saracco GM. Performance of protein induced by vitamin K absence or antagonist-II assessed by chemiluminescence enzyme immunoassay for hepatocellular carcinoma detection: a meta-analysis. Scand J Gastroenterol. 2018 Jun;53(6):734-740. doi: 10.1080/00365521.2018.1459824. Epub 2018 Apr 18. PMID 29667463
- [Background] Choi JY, Jung SW, Kim HY, Kim M, Kim Y, Kim DG, Oh EJ. Diagnostic value of AFP-L3 and PIVKA-II in hepatocellular carcinoma according to total-AFP. World J Gastroenterol. 2013 Jan 21;19(3):339-46. doi: 10.3748/wjg.v19.i3.339. PMID 23372355
- [Background] D'Ambrosio R, Colombo M. Should surveillance for liver cancer be modified in hepatitis C patients after treatment-related cirrhosis regression? Liver Int. 2016 Jun;36(6):783-90. doi: 10.1111/liv.13106. Epub 2016 Mar 24. PMID 26936383
- [Background] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846